CLINICAL TRIAL: NCT02023723
Title: Evaluation of Energy Drink Consumption on ECG and Hemodynamic Parameters in Young Healthy Volunteers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: David Grant U.S. Air Force Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: FDG20130042H
Record Dates: First submitted 2013-12-24; First posted 2013-12-30 (Estimated); Last update posted 2020-04-22 (Actual); Status verified 2020-04

CONDITIONS: Hemodynamic Effects of Energy Drink; Electrocardiograph Effects of Energy Drinks
Keywords: Energy Drink; Electrocardiograph; Hemodynamic
MeSH Terms: interventions — Energy Drinks

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Energy Drink (Experimental): 16oz original flavor energy drink consume 2 -16oz energy drinks within 60 minutes
  Interventions: Dietary Supplement: Energy Drink; Dietary Supplement: Active Control
- Active Control (Active Comparator): 16oz control drink: Caffeine 160mg, Sucrose 115g consume 2 - 16oz drinks within 60 minutes
  Interventions: Dietary Supplement: Energy Drink; Dietary Supplement: Active Control

INTERVENTIONS:
Dietary Supplement: Energy Drink — 16oz energy drinks - 2 consumed within 60 minutes
Dietary Supplement: Active Control — 16oz control drink: Caffeine 160mg, Sucrose 115g consume 2 - 16oz drinks within 60 minutes

SUMMARY:
This study is designed as a safety assessment to determine the cardiac and hemodynamic effects of overuse of energy drinks in healthy individuals through ECG, heart rate (HR) and blood pressure measurements. It will evaluate the use of a consumer available product that is classified as a dietary supplement by the FDA.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female, active duty military service members or DoD beneficiaries, who are eligible to receive care at DGMC.
* Ages 18-40 years old
* Participants must be willing to refrain from caffeine and energy drink use 48 hours prior to study days 1 and 8. They must also refrain from consuming additional caffeine or energy drinks during the 24-hour observation time on days 1-2 and 8-9.

Exclusion Criteria:

* Cardiovascular risk factors: Heart rhythm other than normal sinus, history of atrial or ventricular arrhythmia, family history of premature sudden cardiac death before the age of 60, left ventricular hypertrophy, atherosclerosis, hypertension, palpitations, T-wave abnormalities, baseline corrected QT (QTc) interval greater than 440 milliseconds(ms). This will be determined on the ECG obtained during initial screening appointment, and reviewed by cardiologist and through the questionnaire responses of the participant.
* Blood pressure at initial screening appointment or at baseline on study Day 1 greater than 140/90
* Presence of any known medical condition, confirmed through participant interview. Examples of these are:
* Hypertension
* Thyroid disease
* Type 1 or 2 diabetes mellitus
* Recurrent headaches
* Depression, currently receiving treatment (due to possible drug interactions)
* Any psychiatric condition or neurological disorder
* History of alcohol or drug abuse in the previous 5 years
* Ever been diagnosed or told they have or had renal or hepatic dysfunction
* Concurrent use of ANY medication taken on a daily basis, to include herbal products or supplements. Daily basis is defined as greater than 2 days per week.
* Pregnant or lactating females will be excluded from participation with urine dipstick tests used to confirm pregnancy (pregnancy test performed before each treatment session, days 1 and 8)
* All non-English speaking / writing subjects and those that do not understand the study or consent process will be excluded from the study due to unavailability of medical qualified translator at all times during the study.
* If the subject refuses to sign the informed consent document or HIPAA Authorization, they will be excluded as well

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2013-12; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
QT/QTc measured on an office ECG | 6 hours over 5 visits

SECONDARY OUTCOMES:
Peripheral Blood pressure | 6 hours with 5 visits
  systolic and diastolic
Central blood pressure | 6 hours over 5 visits
  utilizing an applanation tonometry device
Augmentation Index, pulse wave | 6 hours over 5 visits

CONTACTS AND LOCATIONS:
Overall Officials: Emily Fletcher, PhamD, Principal Investigator — David Grant AF Medical Center
Locations (1):
- David Grant AF Medical Center, Travis Air Force Base, California, United States

REFERENCES:
- [Derived] Fletcher EA, Lacey CS, Aaron M, Kolasa M, Occiano A, Shah SA. Randomized Controlled Trial of High-Volume Energy Drink Versus Caffeine Consumption on ECG and Hemodynamic Parameters. J Am Heart Assoc. 2017 Apr 26;6(5):e004448. doi: 10.1161/JAHA.116.004448. PMID 28446495